CLINICAL TRIAL: NCT04380441
Title: Development of a Quality of Life Decision-Making Model for Older Patients With Acute Myeloid Leukemia
Brief Title: Quality of Life Model for Older Patients With AML
Status: Active, not recruiting | Type: Observational
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Other Study IDs: MCC-20585
Record Dates: First submitted 2020-05-05; First posted 2020-05-08 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: AML, Adult; Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to describe the differences in quality of life (QOL) among newly diagnosed patients diagnosed with acute myeloid leukemia (AML) to help design a patient decision-making QOL model for aligning patients' choice of treatment with what matters the most to them.

ELIGIBILITY:
Inclusion Criteria:

* 60 years of age or older
* Newly diagnosed with pathology-confirmed diagnosis of Acute Myeloid Leukemia
* Within 7 days of starting a new treatment
* Must be able to read and speak English at the 8th grade level

Exclusion Criteria:

* Under 60 years of age
* Other malignancy, dementia, traumatic brain injury or individuals with central nervous system involvement of their leukemia

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of the Malignant Hematology Department or Senior Adult Oncology Division at Moffitt Cancer Center in Tampa, Florida.
Sampling Method: Non-Probability Sample
Enrollment: 206 (Actual)
Dates: Start 2020-07-08 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Difference in Quality of Life score between patients receiving intensive versus non-intensive chemotherapy | At baseline and at 30, 60, 90 and 180 days post treatment
  Difference in Quality of Life between newly diagnosed AML patients 60 years of age and older receiving intensive versus non-intensive chemotherapy. Quality of Life will be measured using the Functional Assessment of Cancer Therapy, Leukemia Version (FACT-Leu), a 44-item self reported leukemia specific questionnaire. The FACT-Leu uses a 0-4 Likert scale, 0=not at all and 4=very much. Positive items receive scores from 0-4 points, and negative items are scored from 4-0 points.The FACT-Leu scores are obtained by summing item responses coded so that larger scores indicate better QOL. The leukemia subscale has been validated. A meaningful clinical change for the FACT-Leu is a 13-17 point difference out of a maximum score of 176.
Difference in Quality of Life score between patients with varying disease characteristics | At baseline and at 30, 60, 90 and 180 days post treatment
  Difference in Quality of Life score between patients with varying disease characteristics such as age, performance status, functional status, comorbidity, fatigue, symptoms, blast percentage, transfusion dependence and cytogenic risk group. Quality of Life will be measured using the Functional Assessment of Cancer Therapy, Leukemia Version (FACT-Leu), a 44-item self reported leukemia specific questionnaire. The FACT-Leu uses a 0-4 Likert scale, 0=not at all and 4=very much. Positive items receive scores from 0-4 points, and negative items are scored from 4-0 points. The FACT-Leu scores are obtained by summing item responses coded so that larger scores indicate better QOL. The leukemia subscale has been validated. A meaningful clinical change for the FACT-Leu is a 13-17 point difference out of a maximum score of 176.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Tinsley, PhD, APRN, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Informed Consent Form (2022-07-21): https://cdn.clinicaltrials.gov/large-docs/41/NCT04380441/ICF_000.pdf